CLINICAL TRIAL: NCT06249802
Title: Beta-blockade in Unruptured Intracranial Aneurysm
Acronym: BBLURAN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Collaborators: University Hospital in Krakow (Other)
Responsible Party: Principal Investigator, Jerzy Gąsowski, Prof., Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BBLURAN-CMUJ-14062023
Record Dates: First submitted 2024-01-06; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Intracranial Aneurysm
Keywords: beta-blocker; intracranial aneurysm; rupture prevention; hemodynamic analysis; randomized clinical trial
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Nebivolol

STUDY DESIGN:
Intervention Model Description: Patient recruitment into study will be continuous during first three years of project duration. Two arms will be created - receiving nebivolol or placebo. Dosage of nebivolol will be determined based on blood pressure and heart rate. The investigators aim to enroll a total of 100 patients - 50 for β-blocker treatment arm and 50 for placebo arm. At baseline, included patients will undergo detailed clinical examination, MRI to assess aneurysm morphology and wall, as well as vascular Doppler ultrasound to provide boundary condition for computer modelling. During first 6 months of trial, monthly control visits for each patient will be established, during which they will undergo physical examination. After 6 and 12 months all examinations will be repeated. Further follow-up will then be adopted.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nebivolol arm (Experimental): Patients randomly assigned to receive active treatment with escalating doses of nebivolol.
  Interventions: Drug: Nebivolol
- Placebo arm (Placebo Comparator): Patients randomly assigned to receive matching placebo tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nebivolol — 12-month intake of medication
  Arms: Nebivolol arm
Drug: Placebo — 12-month intake of matching placebo
  Arms: Placebo arm

SUMMARY:
Subarachnoid haemorrhage is a devastating type of stroke, with high mortality and morbidity rate. In approximately 85% of cases, it is caused by an intracranial aneurysm rupture. Majority of patients with diagnosed intracranial aneurysm are eligible for interventional treatment, however, some patients are managed conservatively. Currently, the only recommendations for patients with conservatively managed intracranial aneurysms, are routine imaging follow-ups and minimization of rupture risk factors. There are no medications proven to decrease risk of aneurysm rupture, that might be prescribed to such patients. In preliminary study the investigators found that patients with intracranial aneurysms who took β-blockers had significantly smaller aneurysm rupture rate and dome size, as well as more favorable hemodynamic parameters. No other antihypertensive drugs showed similar associations. Therefore, in this project the investigators aim to further analyze the impact of β-blocker intake on fate of intracranial aneurysm and find possible explanations for its protective role. The investigators aim to perform a randomised, double-blind, placebo-controlled clinical trial. One hundred patients with unruptured intracranial aneurysm, , qualified to conservative management will be enrolled. Two arms (50 patients each) will be receiving nebivolol or matching placebo. Treatment in each arm will last 12 months. The following examinations will be performed at baseline and at 6 and 12 months: clinical assessment, angio-MRI with vessel wall imaging, Doppler ultrasound to extract blood flow waveforms from Internal Carotid Artery, Vertebral Artery Middle Cerebral Artery, Anterior Cerebral Artery and Posterior Cerebral Artery, as well as blood samples. Based on the results the investigators will assess changes in aneurysm size and wall contrast enhancement. The investigators will also analyze levels of possible aneurysm growth biomarkers in peripheral blood. Additionally, the investigators will prepare three-dimensional models of the artery harbouring aneurysm and perform patient-specific computer modelling of blood flow through such artery to assess hemodynamic parameters of aneurysm dome. All obtained measurements will be compared at baseline and at 6 and 12 months. The investigators hypothesize that, in comparison to the placebo group, β-blocker therapy in patients with unruptured intracranial aneurysm will contribute to favorable changes in hemodynamic parameters of aneurysm dome, decrease wall degradation process and prevent from aneurysm growth.

ELIGIBILITY:
Inclusion Criteria:

* freshly (within 12 months) diagnosed unruptured intracranial aneurysm, non-eligible for surgical or endovascular treatment
* age > 18 years
* informed consent

Exclusion Criteria:

* contraindications to β-blockers intake
* previous SAH
* intake of β-blocker currently or in the past
* presence of other intracranial pathology
* history of surgical or endovascular aneurysm treatment
* contraindications for contrast-enhancement MRI examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial aneurysm growth | 12 months
  Any increase in size of intracranial aneurysm assessed by radiology specialist based on Magnetic Resonance Angiography.
Intracranial aneurysm rupture | 12 months
  Fatal or non-fatal intracranial aneurysm rupture. Outcome will be determined based on presence of subarachnoid hemorrhage on head Computer Tomography (performed in case on any symptoms).

SECONDARY OUTCOMES:
All-cause mortality | 12 months
  Death of any cause
Change in aneurysmal hemodynamic parameters | 12 months
  5% increase or decrease (relative to measurement at baseline) of one or more following parameters:
  * dome fraction very high Oscillatory Shear Index (defined as percentage of aneurysm dome with Oscillatory Shear Index higher than 0.2)
  * dome fraction of very low Wall Shear Stress (defined as percentage of aneurysm dome with Wall Shear Stress lower than 0.5)
  * Surface Vortex Fraction (defined as as percentage of flow with positive Q-criterion in small layer near aneurysm wall) All parameters will be determined based on computer modelling of blood flow in aneurysm dome.
Change in aneurysm growth biomarkers | 12 months
  Any change in serum levels of one or more biomarkers: IL-1,IL-6, IL-15, TGF- β and MCP-1.

OTHER OUTCOMES:
5-year all-cause mortality, intracranial aneurysm rupture or necessity of neurosurgical intervention | 5 years
  Yearly follow-up for all-cause mortality or intracranial aneurysm rupture or neurosurgical intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital in Krakow, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided